CLINICAL TRIAL: NCT00948545
Title: Autonomic Nervous System Function and Novel Determinants of Glucose Homeostasis Following Bariatric Surgery
Brief Title: Autonomic Nervous System Function Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: American Society for Metabolic and Bariatric Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: 29092
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Bariatric Surgery
Keywords: Autonomic nervous system; Bariatric surgery; Observational study for individuals having bariatric surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Observing individuals pre and post bariatric surgery
  Interventions: Other: Observational study - there is no intervention

INTERVENTIONS:
Other: Observational study - there is no intervention — Observational study - there is no intervention

SUMMARY:
In the proposed study, the investigators will explore three specific aims. First, the investigators will examine cross-sectionally the association of obesity on sympathetic, parasympathetic, and sympathetic/ parasympathetic nerve fiber balance. In addition, the investigators will determine the relationship of the ANS and osteocalcin. Osteocalcin will be measured before and after a mixed meal tolerance test.

In the second specific aim, the investigators will prospectively follow-up these individuals (n=30) following bariatric surgery. The effect of weight loss on measures of the ANS and osteocalcin will be examined 6 months following surgery with participants serving as their own control, pre- and post-surgical intervention.

Thirdly, the investigators will address whether the effect of weight loss on the ANS and osteocalcin differ between those who had a history of diabetes at baseline versus those with no history of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 - 60 years old.
2. Individuals with a BMI > 35 kg/m2.
3. Patients that have enrolled in a program to undergo weight loss by Roux-en-Y gastric bypass and having passed the pre-operative clearance program.
4. Individuals with diabetes who are currently being treated with diet, exercise, and/or oral medications will be included.

Exclusion Criteria:

1. Patients that have had previous gastric surgery, including but not limited to pancreobiliary diversion, vertical banded gastroplasty, and jejunoileostomy.
2. Individuals with known coronary artery disease (e.g., post-MI), atrial fibrillation,frequent atrial arrhythmias, frequent ventricular arrhythmias, a pacemaker, or myocardial ischemia.
3. Individuals taking the following medications that may affect the autonomic nervous system: anti- tuberculosis drugs, nitrofurantoin, metronidazole, chloramphenicol,perhexiline maleate, amiodarone, clofibrate, tricyclic antidepressants, phenytoin,methotrexate, barbiturates, neuroleptic drugs, antiparkinsonism drugs, fluoxetine, and nitrated drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals having bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine the association of obesity on sympathetic, parasympathetic, and sympathetic/parasympathetic nerve fiber balance and to determine the relationship of the ANS and osteocalcin. | 2 years

SECONDARY OUTCOMES:
To determine the effect of weight loss on measures of the ANS and determinants of insulin sensitivity (e.g., osteocalcin) 6 months following surgery with participants serving as their own control, pre- and post-surgical intervention. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: M James Lenhard, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States